CLINICAL TRIAL: NCT02958332
Title: Effects of a Videogame-based Program on Women With Lymphedema Secondary to Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-MSV-19-09-2016
Record Dates: First submitted 2016-10-28; First posted 2016-11-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Lymphedema; Breastcancer
Keywords: video games
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- video game program (Experimental): Participants will play video games during 30 min , all along 5 sessions.
  Interventions: Other: video game program

INTERVENTIONS:
Other: video game program — Participants will use the Wii console and the Wii balance board, to play different video games which imply shoulder movements. They will receive 5 individual sessions of 30 minutes.

SUMMARY:
Aims: To demonstrate the effect of a program based on video games as a means to improve abilities and basic skills affected by lymphedema, and its impact on quality of life.

Design: longitudinal, pre-experimental, with pre / post-test and evaluation, assessor blinded study.

Method: Data on shoulder pain and disability, health-related quality of life, strength and articulate activated by the OSS (Oxford Shoulder Score), SPADI (Shoulder Pain and Disability Index), FACT-B + 4 (Functional Assesment of Cancer Therapy Questionnaire for Breast Cancer), respectively goniometry and dynamometry amplitude scales will be collected.

The intervention will be performed with the Wii ™ console and the Wii Balance BoardTM, during 5 individual weekly sessions of 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years
* Have a diagnosis of lymphedema, secondary to breast cancer

Exclusion Criteria:

* Stage 0 or subclinical lymphedema
* Present other shoulder pathology apart from lymphedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Range motion | Pre intervention and one week after having finished the program
Change in strength | Pre intervention and one week after having finished the program
Change in Oxford Shoulder Scale | Pre intervention and one week after having finished the program
Change in Shoulder Pain and Disability Index | Pre intervention and one week after having finished the program

SECONDARY OUTCOMES:
Change in quality of life (FUNCTIONAL ASSESMENT OF CANCER THERAPY QUESTIONNAIRE FOR BREAST CANCER (FACT-B+4) | Pre intervention and one week after having finished the program

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Santamaría-Vázquez, PhD, Principal Investigator — Universidad de Burgos
Locations (1):
- Universidad de Burgos. Facultad de Ciencias de la Salud., Burgos, Spain